CLINICAL TRIAL: NCT00623519
Title: Assessment of Endometrial Changes in Postmenopausal Women With Breast Cancer in Adjuvant Treatment With Anastrozole.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Rosana Cajal, MD - Medical Director, AstraZeneca Spain
Other Study IDs: AST-ANA-2004-01
Record Dates: First submitted 2008-02-06; First posted 2008-02-26 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Breast Cancer
Keywords: Adjuvant postmenopausal breast cancer women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Women with hormone receptor positive breast cancer under adjuvant treatment with Anastrozole

SUMMARY:
To investigate the global incidence of the endometrial changes in postmenopausal women receiving Anastrozole for the adjuvant treatment of hormone receptors positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Provision of Informed Consent
* Resectable breast cancer patients, with histological confirmation
* Patients eligible to receive hormonal adjuvant treatment with Anastrozole
* They are allowed patients treated with adjuvant chemo or radiotherapy concurrently
* Patients previously treated with Tamoxifen that had to withdraw treatment due to other reason than endometrial changes are allowed
* Postmenopausal patients(aged 50 years or over/ without menses in the last months/ FSH level >40UI/L / women under 50 years with FSH levels>40UI/L).
* Women showing progesterone and/or estrogen receptors positive.

Exclusion Criteria:

* Patients with evidence of metastatic disease
* Patients unsuitable to receive the medication according the Anastrozole label
* Patients not giving their Informed Consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical Oncology
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2004-06; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Global incidence of endometrial changes during the adjuvant treatment with Anastrozole | From inclusion to treatment end(5 years duration) measurements will be taken annually, with a further assessment 12 months after end of treatment.

SECONDARY OUTCOMES:
To describe the endometrial changes both clinically(vaginal bleeding) and through the scan. | During the study, at least annually
Histological assessment when indicated(type of hyperplasia) | When applicable
To assess global incidence of endometrial changes in this patient population before taking Anastrozole | During the study
To evaluate type of surgery required for endometrial changes control(hysterectomy rate) | During the study
To assess treatment tolerability | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Rosana Cajal, MD, Study Director — AstraZeneca Spain
Locations (12):
- Spain (12):
  - Research Site, A Coruña
  - Research Site, Granada
  - Research Site, Huelva
  - Research Site, Ibiza Town
  - Research Site, Jerez de la Frontera
  - Research Site, La Rioja
  - Research Site, Lugo
  - Research Site, Mallorca
  - Research Site, Málaga
  - Research Site, Pontevedra
  - Research Site, Santander
  - Research Site, Seville